CLINICAL TRIAL: NCT06653153
Title: A Study of Remternetug Versus Placebo in Early Alzheimer's Disease Participants at Risk for Cognitive and Functional Decline
Brief Title: A Study of Remternetug (LY3372993) in Early Alzheimer's Disease (TRAILRUNNER-ALZ 3)
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 27183; J1G-MC-LAKI (Other: Eli Lilly and Company); 2024-515656-20-00 (EU CTIS Number)
Record Dates: First submitted 2024-10-21; First posted 2024-10-22 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Remternetug (Experimental): Remternetug administered subcutaneously (SC).
  Interventions: Drug: Remternetug
- Placebo (Placebo Comparator): Placebo administered SC.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Remternetug — Administered SC
  Other Names: LY3372993
  Arms: Remternetug
Drug: Placebo — Administered SC
  Arms: Placebo

SUMMARY:
The purpose of this study is to measure the difference in time to developing or worsening memory, thinking, or functional problems due to Alzheimer's disease occurring in participants receiving study drug compared to placebo.

Participation could last up to 255 weeks including screening, a double-blind treatment period, and a double-blind observation period. In addition, eligible participants who receive placebo during the double-blind treatment period may choose to extend their study participation to receive open-label remternetug in an extension period.

ELIGIBILITY:
Inclusion Criteria:

* Have a phosphorylated tau (P-tau) result consistent with the presence of amyloid pathology.
* Have a reliable study partner and backup study partner familiar with overall function and behavior, such as day-to-day activities and cognitive abilities.
* Have adequate literacy, vision, and hearing for neuropsychological testing at screening.
* Have a Mini Mental Status Exam (MMSE) score consistent with no to minimal cognitive impairment.
* Have a Functional Activities Questionnaire (FAQ) score consistent with no to minimal functional impairment.
* If currently receiving medications as symptomatic treatment for AD, dose has been stable for at least 30 days before screening.

Exclusion Criteria:

* Have dementia or significant other neurological disease that can affect cognition.
* Have current serious or unstable illnesses that in the investigator's opinion, could interfere with the analyses of the study.
* Have a history of cancer that, in the investigator's opinion, has a high risk of recurrence.
* Have a history of clinically significant multiple or severe drug allergies, or hypersensitivity reactions.
* Have a clinically important laboratory test result or other abnormality as determined by investigator, prior to randomization, that could be detrimental to the participant or could compromise the study.
* Have any contraindications for magnetic resonance imaging (MRI).
* Have a centrally read MRI that does not meets study entry criteria.

Prior or Current Therapies

* Have ever had prior treatment with a passive anti-amyloid immunotherapy.
* Have received active immunization against Aβ in any other study.

Ages: 55 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1400 (Estimated)
Dates: Start 2024-10-24 (Actual); Primary Completion 2029-04 (Estimated); Study Completion 2030-10 (Estimated)

PRIMARY OUTCOMES:
Time to Clinically Meaningful Progression as Measured by Clinical Dementia Rate Scale (CDR) | Baseline to Time to Event up to Week 255
  Time to clinically meaningful progression as measured by CDR. CDR is a clinician-rated scale that provides an overall assessment of the participant's stage and degree of impairment across the continuum of early Alzheimer's Disease (AD).

SECONDARY OUTCOMES:
Change from Baseline in Clinical Dementia Rate Box Score (SB) | Baseline, Week 255
  Change from baseline in Clinical Dementia Rate Box Score (SB) scores range from 0 to 18, with higher scores indicative of more impairment.
Change from Baseline in Montreal Cognitive Assessment (MoCA) | Baseline, Week 255
  Change from baseline in Montreal Cognitive Assessment (MoCA). Total MoCA score is 0 to 30, with lower scores indicating greater level of impairment.
Change from Baseline in the Category Fluency - Language, Executive Function, Semantic Memory | Baseline, Week 255
  Change from baseline in the Category Fluency - Language, Executive Function, Semantic Memory. The total score reflects the sum of correct responses generated across all categories presented, with higher values indicating better performance.
Change from Baseline in the Continuous Paired Associate Learning (CPAL) | Baseline, Week 255
  Change from baseline in Continuous Paired Associate Learning (CPAL) - Visual episodic memory.
Change from Baseline in International Shopping List Test (ISLT) - Verbal Episodic Mem | Baseline, Week 255
  Change from baseline in the International Shopping List Test (ISLT) - verbal episodic memory.
Change from Baseline in International Daily Symbol Substitution Test-Medicines (iDSSTm) - Complex Attention Memory | Baseline, Week 255
  Change from baseline in the International Daily Symbol Substitution Test-Medicines (iDSSTm) - complex attention memory.
Change from Baseline in Cognitive Function Index (CFI) | Baseline, Week 255
  Change from baseline in the Cognitive Function Index (CFI).
Change from Baseline in Mild Behavioral Impairment Checklist (MBI-C) | Baseline, Week 255
  Change from baseline in the Mild Behavioral Impairment Checklist (MBI-C) The MBI-C total score range is 0 to 102, with higher scores indicating greater impairment.
Change from Baseline in Alzheimer's Disease Cooperative Study (ADCS) Activities of Daily Living - Prevention Instrument (ADCS-ADL-PI) | Baseline, Week 255
  Change from baseline in the Activities of Daily Living - Prevention Instrument total scores range from 0 to 54, with higher scores indicating better performance.
Pharmacokinetics: Serum Concentrations of Remternetug | Baseline through Week 255
  PK: serum concentration of remternetug.
Number of Participants with Treatment Emergent Anti-Drug Antibodies (TE-ADAs) | Baseline through Week 255
  Number of participants with treatment emergent anti-drug antibodies (TE-ADAs).

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 8 AM - 8 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (262):
- United States (123):
  - Parkway Medical Center, Birmingham, Alabama
  - MD First Research - Chandler, Chandler, Arizona
  - Care Access - 801 South Power Road, Mesa, Mesa, Arizona
  - Banner Alzheimer's Institute, Phoenix, Arizona
  - Banner Alzheimer's Institute Tucson, Tucson, Arizona
  - Neuro-Pain Medical Center, Fresno, California
  - Care Access - Huntington Beach, Huntington Beach, California
  - Inglewood Clinical, Inglewood, California
  - Irvine Clinical Research, Irvine, California
  - Healthy Brain Clinic, Long Beach, California
  - Riverside Clinical, Riverside, California
  - Clinical Trials Research, Sacramento, California
  - Artemis Institute for Clinical Research, San Diego, California
  - Sharp Neurocognitive Research Center, San Diego, California
  - Ray Dolby Brain Health Center, San Francisco, California
  - The Neuron Clinic - San Marcos, San Marcos, California
  - Syrentis Clinical Research, Santa Ana, California
  - Providence Medical Foundation, Santa Rosa, California
  - California Neuroscience Research, LLC, Sherman Oaks, California
  - Care Access - Aurora, Aurora, Colorado
  - Mountain Neurological Research Center, Basalt, Colorado
  - Alpine Clinical Research Center, Boulder, Colorado
  - CenExel Rocky Mountain Clinical Research, Englewood, Colorado
  - Invicro, New Haven, Connecticut
  - Ki Health Partners, LLc, dba New England Institute for Clinical Research, Stamford, Connecticut
  - JEM Research Institute, Atlantis, Florida
  - VIN - Aventura, Aventura, Florida
  - Bradenton Research Center, Inc., Bradenton, Florida
  - K2 Medical Research WINTER GARDEN, Clermont, Florida
  - TecTum Research, Davie, Florida
  - Brain Matters Research, Delray Beach, Florida
  - Neuropsychiatric Research Center of Southwest Florida, Fort Myers, Florida
  - Indago Research & Health Center, Inc, Hialeah, Florida
  - K2 MEDICAL Research THE VILLAGES, Lady Lake, Florida
  - ClinCloud, Maitland, Florida
  - K2 Medical Research ORLANDO, Maitland, Florida
  - ClinCloud, Melbourne, Florida
  - Merritt Island Medical Research, LLC, Merritt Island, Florida
  - VIN-Andrew Lerman, Miami, Florida
  - New Age Medical Research Corporation, Miami, Florida
  - Adult Medicine of Lake County, Inc., Mt. Dora, Florida
  - Aqualane Clinical Research, Naples, Florida
  - Suncoast Clinical Research, Inc., New Port Richey, Florida
  - Renstar Medical Research, Ocala, Florida
  - Charter Research - Winter Park, Orlando, Florida
  - AdventHealth Orlando, Orlando, Florida
  - Emerald Coast Neurology - Airport Boulevard, Pensacola, Florida
  - Progressive Medical Research, Port Orange, Florida
  - Alzheimer's Research and Treatment Center, Stuart, Florida
  - Axiom Brain Health LLC, Tampa, Florida
  - Stedman Clinical Trials, Tampa, Florida
  - Care Access - Tampa, Tampa, Florida
  - Charter Research - Lady Lake, The Villages, Florida
  - Alzheimer's Research and Treatment Center, Wellington, Florida
  - Palm Beach Neurology, West Palm Beach, Florida
  - Conquest Research, Winter Park, Florida
  - Columbus Memory Center, LLC, Columbus, Georgia
  - Care Access - Decatur, Decatur, Georgia
  - Center for Advanced Research & Education, Gainesville, Georgia
  - North Georgia Clinical Research, Woodstock, Georgia
  - Northwest Clinical Trials, Boise, Idaho
  - Care Access - Arlington Heights, Arlington Heights, Illinois
  - Re:Cognition Health - Chicago, Chicago, Illinois
  - Great Lakes Clinical Trials - Andersonville, Chicago, Illinois
  - Alexian Brothers Medical Center, Elk Grove Village, Illinois
  - Care Access - South Indianapolis, Indianapolis, Indiana
  - Josephson Wallack Munshower Neurology, PC, Indianapolis, Indiana
  - Cedar Valley Medical Specialists, Waterloo, Iowa
  - Cotton O'Neil Clinical Research Center, Topeka, Kansas
  - Care Access - Lake Charles (Bayou Pines), Lake Charles, Louisiana
  - Tandem Clinical Research, Marrero, Louisiana
  - Acadia Hospital, Bangor, Maine
  - Care Access - Baltimore, Baltimore, Maryland
  - Adams Clinical Boston, Boston, Massachusetts
  - Boston Clinical Trials, Boston, Massachusetts
  - Boston Center for Memory, Newton, Massachusetts
  - Care Access - Quincy, Quincy, Massachusetts
  - MedVadis Research Corporation, Waltham, Massachusetts
  - Adams Clinical Watertown, Watertown, Massachusetts
  - Revival Research Institute, LLC, Dearborn, Michigan
  - QUEST Research Institute, Farmington Hills, Michigan
  - HealthPartners Neuroscience Center, Saint Paul, Minnesota
  - Private Practice - Dr. Ronald Louis Schwartz, Hattiesburg, Mississippi
  - Citizens Memorial Hospital District, Bolivar, Missouri
  - Clinical Research Professionals, Chesterfield, Missouri
  - University Of Nebraska Medical Center, Omaha, Nebraska
  - Vector Clinical Trials, Las Vegas, Nevada
  - Care Access - Hoboken, Hoboken, New Jersey
  - The Cognitive and Research Center of New Jersey - Ridgewood, Ridgewood, New Jersey
  - The Cognitive and Research Center of New Jersey, Springfield, New Jersey
  - Advanced Memory Research Institute of New Jersey, Toms River, New Jersey
  - IMA Clinical Research, Albuquerque, New Mexico
  - Care Access - Charlotte, Charlotte, North Carolina
  - Medication Management, Greensboro, North Carolina
  - Monroe Biomedical Research, Monroe, North Carolina
  - Care Access - Lima, Lima, Ohio
  - North Star Medical Research, Middleburg Heights, Ohio
  - Summit Headlands, Portland, Oregon
  - Clinical Research of Philadelphia, Philadelphia, Pennsylvania
  - Keystone Clinical Studies, Plymouth Meeting, Pennsylvania
  - Rhode Island Mood & Memory Research Institute, East Providence, Rhode Island
  - Butler Hospital, Providence, Rhode Island
  - Tribe Clinical Research, LLC- Greenville, Greenville, South Carolina
  - Palmetto Clinical Research, Summerville, South Carolina
  - Neurology Clinic, P.C., Cordova, Tennessee
  - Genesis Neuroscience Clinic, Knoxville, Tennessee
  - Senior Adults Specialty Research, Austin, Texas
  - Gadolin Research, Beaumont, Texas
  - Kerwin Medical Center - Oak Cliff, Dallas, Texas
  - Kerwin Medical Center, Dallas, Texas
  - Care Access - Georgetown, Georgetown, Texas
  - Care Access - Houston, Houston, Texas
  - The University of Texas Health Science Center at Houston, Houston, Texas
  - Next Level Urgent Care, Houston, Texas
  - El Faro Health and Therapeutics, Rio Grande City, Texas
  - Central Texas Neurology Consultants, PA, Round Rock, Texas
  - IMA Clinical Research San Antonio, San Antonio, Texas
  - Consano Clinical Research, LLC, Shavano Park, Texas
  - Care Access - Arlington 2, Arlington, Virginia
  - Re:Cognition Health, Fairfax, Virginia
  - Eastern Virginia Medical School (EVMS) Medical Group, Norfolk, Virginia
  - Northwest Clinical Research Center, Bellevue, Washington
  - Rainier Clinical Research Center, Renton, Washington
- Australia (16):
  - USC Clinical Trials Sunshine Coast, Birtinya
  - Emeritus Research, Botany
  - Box Hill Hospital, Box Hill
  - Emeritus Research, Camberwell
  - GenesisCare - Maitland, East Maitland
  - The University of Queensland, Herston
  - Ipswich Hospital, Ipswich
  - Austin Health, Ivanhoe
  - Southern Neurology, Kogarah
  - KARA Institute for Neurological Diseases, Macquarie Park
  - HammondCare, Malvern
  - Fusion Clinical Research, Norwood
  - The Royal Melbourne Hospital, Parkville
  - USC Clinical Trials Brisbane (South Bank), South Brisbane
  - St Vincent's Hospital, Sydney
  - The Queen Elizabeth Hospital, Woodville
- Canada (17):
  - Ecogene-21 - Cmas, Chicoutimi
  - MoCA Research and Innovation Inc., Greenfield Park
  - OCT Research ULC, Kelowna
  - Alpha Recherche Clinique - Lévis, Lévis
  - Clinique Mémoire de Montréal, Montreal
  - Genge Partners, Montreal
  - Ottawa Memory Clinic, Ottawa
  - Kawartha Centre - Redefining Healthy Aging, Peterborough
  - Alpha Recherche Clinique, Québec
  - ALPHA Recherche Clinique, Québec
  - Bluewater Clinical Research Group Inc., Sarnia
  - Q&T Research Sherbrooke Inc., Sherbrooke
  - Toronto Memory Program, Toronto
  - Sunnybrook Research Institute, Toronto
  - Baycrest Health Sciences, Toronto
  - Diex Recherche Inc. Division Victoriaville, Victoriaville
  - The Medical Arts Health Research Group - West Vancouver, West Vancouver
- China (29):
  - Beijing Tiantan Hospital Affiliated to Capital Medical University, Beijing
  - Beijing Anding Hospital - Affiliated Capital University of Medical Science, Beijing
  - The First Hospital of Jilin University, Changchun
  - Xiangya Hospital Central South University, Changsha
  - Sichuan Provincial People's Hospital, Chengdu
  - Guangdong Provincial People's Hospital, Guangzhou
  - Guangzhou First People's Hospital, Guangzhou
  - Guangzhou Medical University 2nd Hospital, Guangzhou
  - Zhujiang Hospital, Guangzhou
  - Anhui Provincial Hospital, Hefei
  - Jinan Central Hospital, Jinan
  - The First Affiliated Hospital of Henan University of Science &Technology, Luoyang
  - The Second Affiliated Hospital of Nanchang University, Nanchang
  - The First Affiliated Hospital of Nanchang University, Nanchang
  - Nanjing Brain Hospital, Nanjing
  - Sir Run Run Hospital of Nanjing Medical University, Nanjing
  - Shanghai Sixth People's Hospital, Shanghai
  - Huashan Hospital, Fudan University, Shanghai
  - Renji Hospital Shanghai Jiao Tong University School of Medicine, Shanghai
  - Pudong New Area People's Hospital Shanghai, Shanghai
  - The First Hospital of Hebei Medical University, Shijiazhuang
  - The Second Affiliated Hospital of Soochow University, Suzhou
  - Tianjin Medical University General Hospital, Tianjin
  - Shaanxi provincial people's hospital, Xi'an
  - The First Affiliated Hospital of Xi'an Medical University, Xi'an
  - Xianyang Hospital of Yan'an University, Xianyang
  - The Affiliated Hospital of Xuzhou Medical College, Xuzhou
  - Xuzhou Central Hospital, Xuzhou
  - Zigong First People's Hospital, Zigong
- Japan (27):
  - The University of Tokyo Hospital, Bunkyō City
  - Medical Corporation Chiseikai Tokyo Center Clinic, Chūōku
  - Tokyo-Eki Center-building Clinic, Chūōku
  - Fukuwa Clinic, Chūōku
  - Tokyo Asbo Clinic, Chūōku
  - Kawashima Neurology Clinic, Fujisawa
  - UNB Sumiyoshi Jinjamae Clinic, Fukuoka
  - Boocs Clinic Fukuoka, Fukuoka
  - P-One Clinic, Hachiōji
  - Hyogo Prefectural Harima-Himeji General Medical Center, Himeji
  - Saiseikai Imabari Hospital, Imabari
  - Kobe University Hospital, Kobe
  - Showa General Hospital, Kodaira
  - Tatsuoka Neurology Clinic, Kyoto
  - Sakurazaka Clinic SophyAnce, Minatoku
  - Iwata Neurosurgery Clinic, Osaka
  - National Center for Geriatrics and Gerontology, Ōbu
  - Kanto Central Hospital, Setagaya-ku
  - Samoncho Clinic, Shinjuku
  - Clinical Research Hospital Tokyo, Shinjuku-ku
  - Heishinkai Medical Group ToCROM Clinic, Shinjuku-ku
  - Higashi Shinjuku Clinic, Shinjuku-ku
  - Medical Corporation Heishinkai OCROM Clinic, Suita-shi
  - Tokyo Metropolitan Geriatric Hospital, tabashi City
  - Tachikawa Hospital, Tachikawa
  - Takatsuki Hospital, Takatsuki-shi
  - Wako Hospital, Wako
- Puerto Rico (4):
  - SCB Research Center, Bayamón
  - Caribbean Medical Research Center, San Juan
  - INSPIRA Clinical Research, San Juan
  - Instituto De Neurologia Dra. Ivonne Fraga, San Juan
- South Korea (17):
  - Pusan National University Hospital, Busan
  - Chungbuk National University Hospital, Cheongju-si
  - Gangnam Severance Hospital, Yonsei University Health System, Gangnam-gu
  - Ewha Womans University Seoul Hospital, Gangseo-gu
  - Chonnam National University Hospital, Gwangju
  - Inha University Hospital, Incheon
  - Jeju National University Hospital, Jeju City
  - Gachon University Gil Medical Center, Namdong-gu
  - Seoul National University Bundang Hospital, Seongnam
  - Seoul National University Hospital, Seoul
  - Hanyang University Seoul Hospital, Seoul
  - Konkuk University Medical Center, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - The Catholic Univ. of Korea Seoul St. Mary's Hospital, Seoul
  - Ajou University Hospital, Suwon
  - Wonju Severance Christian Hospital, Wŏnju
- Spain (7):
  - Barcelonabeta Brain Research Center, Barcelona
  - Fundació ACE, Barcelona
  - Hospital Clínic de Barcelona, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Universitario Quironsalud Madrid, Pozuelo de Alarcón
  - Policlinica Gipuzkoa, San Sebastián
  - Hospital Victoria Eugenia, Seville
- Taiwan (10):
  - Changhua Christian Hospital, Changhua County
  - National Taiwan University Hospital Yun-Lin Branch Dou-Liou Region, Douliu
  - Chang Gung Memorial Hospital at Kaohsiung, Kaohsiung Niao Sung Dist
  - Taipei Medical University Shuang Ho Hospital, New Taipei City
  - New Taipei Municipal TuCheng Hospital, New Taipei City
  - China Medical University Hospital, Taichung
  - Taichung Veterans General Hospital, Taichung
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Chang Gung Medical Foundation-Linkou Branch, Taoyuan District
- United Kingdom (12):
  - ReMind UK, Bath
  - Re:Cognition Health - Birmingham, Birmingham
  - Layton Medical Centre, Blackpool
  - Scottish Brain Sciences, Edinburgh
  - St Pancras Clinical Research, London
  - NIHR Manchester Clinical Research Facility, Manchester
  - NeuroClin, Motherwell
  - Roborough Surgery, Plymouth
  - Homecroft Surgery, Redruth
  - Abbeywell Surgery, Romsey
  - Moorgreen Hospital, Southampton
  - Marine Lake Medical Practice, West Kirby

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: http://vivli.org/